CLINICAL TRIAL: NCT01462253
Title: "A Phase II Study With a Sequential Clofarabine-cyclophosphamide Combination Schedule as Salvage Therapy for Refractory and Relapsed Acute Lymphoblastic Leukemia (ALL) in Adult Patients"
Brief Title: Clofarabine-cyclophosphamide as Salvage Therapy for Refractory and Relapsed Acute Lymphoblastic Leukemia (ALL) Adults
Acronym: LAL1610
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL1610
Record Dates: First submitted 2011-10-21; First posted 2011-10-31 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Adult patients; Refractory; Relapsed; clofarabine; cyclophosphamide; refractory and relapsed acute lymphoblastic leukemia; ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Clofarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clofarabine, Cyclophosphamide (Experimental): Clofarabine concentrate for solution for infusion should be filtered using a 0.2 micron filter and diluted to a final concentration between 0.15 mg/mL and 0.4 mg/mL with 0.9% sodium chloride injection USP or European Pharmacopeia (EP) normal saline (NS), or 5% dextrose injection (D5W) USP or EP prior to infusion.
  Cyclophosphamide should be prepared for parenteral use by adding 0.9% sterile sodium chloride solution. Solutions of cyclophosphamide may be injected intravenously without further dilution or may be infused following further dilution: Dextrose Injection, USP (5% dextrose), Dextrose and Sodium Chloride Injection, USP (5% dextrose and 0.9% sterile sodium chloride), 5% Dextrose and Ringer's Injection.
  Interventions: Drug: Clofarabine, Cyclophosphamide

INTERVENTIONS:
Drug: Clofarabine, Cyclophosphamide — The proposed treatment schedule consists of a combination of Clofarabine plus Cyclophosphamide administered over 5 consecutive days (Treatment scheme).

SUMMARY:
This is a multicentric, prospective pilot trial testing a Clofarabine-Cyclophosphamide combination to treat refractory and first bone marrow relapse adult ALL, for the achievement of a complete remission (CR) and the concurrent evaluation of biological response in ALL cells (minimal residual disease, apoptosis and DNA cell damage, pharmacogenomics).

DETAILED DESCRIPTION:
The proposed treatment schedule consists of a combination of Clofarabine plus Cyclophosphamide administered over 5 consecutive days (Treatment scheme). This is an open, nonrandomized prospective phase II trial aimed to evaluating (1) activity of this combination in terms of CR rate.

* STEP 1. All eligible patients will be screened for the availability of an HLA-matched or partially mismatched compatible HSCT donor, of both family related - or unrelated type (early activation required), including cord blood and haploidentical siblings. Moreover, pre-treatment investigation will include collection and storage of patient ALL cells for specific biological studies relating to sensitivity and response to study chemotherapeutic combination.
* STEP 2. Cycle 1 will be applied to all eligible patients once all enrollment criteria are confirmed.
* STEP 3. After cycle 1, response will be evaluated.
* STEP 4. After remission induction cycle 1, only responsive patients (CR or PR, see below for definitions) could be given cycle 2, according to the opinion of the responsible physician and with a minimum intercycle interval of 4 weeks from day 1 of cycle 1. All NR patients will be declared off study and will not be given a second course with study combination. The suggested treatment following cycle 2 (or cycle 1 if cycle 2 is omitted) is HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to IGH/EU/GCP and national local laws.
* Age 18-60 years.
* ALL with B-/T-precursor phenotype refractory to first line therapy.
* ALL with B-/T-precursor phenotype 1st isolated bone marrow relapse, occurring < 24 months from the achievement of first CR, after chemotherapy or hematopoietic stem-cell transplantation (HSCT) defined as follows:

  * ≥ 5% leukemic blasts in the bone marrow not attributable to another cause (e.g. marrow regeneration); if there are no circulating blasts and the bone marrow contain 5-20% leukemic blasts, a repeat bone marrow performed at least a week later is necessary to confirm relapse.
* ECOG performance status 0-2 or reversible ECOG 3 score following intensive care of complications.
* Adequate hepatic and renal function, unless considered due to organ leukemic involvement:

  * Serum creatinine <1.5 mg/dl; if serum creatinine >1.5 mg/dl, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female), x (1.212) if patient is black.
  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN).
  * Aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2.5 x ULN.
  * Alkaline phosphatase ≤ 2.5 x ULN.

Exclusion Criteria:

* Prior exposure to Clofarabine or, in primary refractory patients only, to Cyclophosphamide during induction courses.
* Patients relapsed > 24 months from first CR. - Philadelphia chromosome-positive (Ph+) ALL.
* Diagnosis of Burkitt-type/B-ALL, or B-/T-lymphoblastic lymphoma with < 25% bone marrow involvement.
* Concurrent or isolated central nervous system (CNS) relapse.
* Pre-existing, uncontrolled pathology such as cardiac disease (congestive/ischemic, acute myocardial infarction within the past 3 months, untreatable arrythmias, NYHA classes III and IV).
* Severe neurological or psychiatric disorder that impairs the patient's ability to understand and sign the informed consent, or to cope with the intended treatment plan.
* Active uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* HIV positive serology or active hepatitis infection. - Concurrent diagnosis of active cancer requiring concurrent chemotherapy and/or radiotherapy, and/or with life expectancy < 1 year.
* Patients who are pregnant or adults of reproductive potential not employing an effective method of birth control (women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of Clofarabine-Cyclophosphamide). Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-10; Primary Completion 2017-03-11 (Actual); Study Completion 2017-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato BASSAN, Pr., Principal Investigator — U.O. di Ematologia- Ospedale dell'Angelo - Mestre
Locations (27):
- Italy (27):
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - Divisione di Ematologia - Ospedali Riuniti, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Sanitaria di Bolzano - Ospedale Centrale - Ematologia e Centro TMO, Bolzano
  - Sezione di Ematologia e Trapianti Spedali Civili, Brescia
  - Azienda ASL di Cagliari, Cagliari
  - Ospedale Santa Croce Divisione di Ematologia Cuneo, Cuneo
  - Policlinico di Careggi, Università delgi studi di Firenze, Florence
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - U.O. di Ematologia- Ospedale dell'Angelo - Mestre, Mestre
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - UO Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - N. Osp. divisione di Ematologia "S.Gerardo dei Tintori", Monza
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale Cervello, Palermo
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Calabria Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Umberto I di Roma - Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - SCDO Ematologia 2 AOU Giovanni Battista, Torino

REFERENCES:
- See also: GIMEMA Foundation Website — http://www.gimema.it/en/index.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Clofarabine + Cyclophosphamide: Patients received a maximum of two consecutive cycles of Clofarabine-Cyclophosphamide, at an intercycle interval of 28 days or greater, according to tolerability and clinical status.
  Cycle 2 was only administered to patients obtaining at least a partial response (PR) after cycle 1.
Period: Overall Study
Arm/Group | Clofarabine + Cyclophosphamide
Started | 35
Completed | 27
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: Years] | 38.7 [20.5 to 59.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 27
Patient status - relapsed [Number; unit: participants] | 25
Patient status - refractory [Number; unit: participants] | 2
White Blood Cells (WBC) [Median (Full Range); unit: cells/microliter] | 5670.0 [104.9 to 55000.0]
Platelets count [Median (Full Range); unit: cells/microliter] | 105000.0 [14000.0 to 270000.0]

OUTCOME MEASURES:

1. Primary Outcome: The Primary End-point is the Number of Patients in CR After Induction Therapy.
Description: Disappearance of any clinical and laboratoristic sign of ALL. The patient must be transfusion-free with neutrophils >1.0 x109/L and platelets >100 x109/L. BM examination must show absence or reduction of blast cell content (< 5%, none of which obviously leukemic), with cellularity in the normal or slightly hypocellular range and with evidence of trilineage hemopoiesis. BM is examined on day 28 from start of chemotherapy cycle 1, or later as clinically indicated in ill/cytopenic patients, and after cycle 2 in patients with PR proceeding to this treatment.
Time Frame: At day +28 from start of chemotherapy cycle 1 and after cycle 2 in pts with PR
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 27
Participants | 9

2. Secondary Outcome: Number of Participants With Toxicity of Grade 2 or Greater
Description: Referring to CTCAE (Common Toxicity Criteria Events), version 4.0
Time Frame: At 13 months from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 27
Participants | 10

3. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD) Response in Remission.
Time Frame: At week 10, 16 and 22 from start of treatment and the, every three months till study completion
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 10
Participants | 1

4. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival (DFS) at 1 year, defined as the time interval between the evaluation of CR and relapse of the disease or death in first CR; patients still alive, in first CR, will be censored at the time of the last follow-up. In this case, the DFS curve will be truncated at 1 year
Time Frame: At one year from completion of chemotherapy
Population: Disease-free survival was estimated in CR patients (n=16) from date of first CR to date of death, relapse or last follow-up.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 16
Percentage of patients | 31.25 [17.3 to 69.7]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) at 1 year; defined as the time interval between inclusion and death for any cause; patients still alive will be censored at the time of the last follow-up. In this case, the OS curve will be truncated at 1 year.
Time Frame: At one year from therapy completion.
Population: Overall survival was estimated from date of informed consent to date of death or last follow-up.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 27
Percentage of patients | 28.6 [15.3 to 53.3]

6. Secondary Outcome: Cumulative Incidence of Relapse (CIR)
Description: Cumulative incidence of relapse (CIR) at 1 year, it will be calculated from the date of achievement of the first CR, using the cumulative incidence method, considering death in CR as a competing risk. Patients still alive, without a date of relapse, will be censored at the time of the last follow-up. In this case, the CIR curve will be truncated at 1 year.
Time Frame: At one year from therapy completion.
Population: Cumulative incidence of relapse was estimated only in CR patients (n=16) from date of first CR to date of death, relapse or last follow-up; considering death in CR as a competing risk.
  Median CIR not yet reached.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Clofarabine + Cyclophosphamide
Number analyzed (Participants) | 16
Percentage of patients | 31.25 [10.774 to 54.485]

ADVERSE EVENTS:
Time Frame: 54 months from study entry
Arm/Group | Clofarabine + Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 4/27
Serious Adverse Events (participants affected / at risk) | 7/27
Other Adverse Events (participants affected / at risk) | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Cyclophosphamide (N=27)
Septic shock (Infections and infestations) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 1 (2)
Pneumonitis (Infections and infestations) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Cyclophosphamide (N=27)
Vena cava thrombois (Vascular disorders) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 3 (5)
Bronchopneumonia (Infections and infestations) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 3 (3)
Nephropathy toxic (Renal and urinary disorders) | 1 (1)
Neurological toxicity (Nervous system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2012-01-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT01462253/SAP_000.pdf
  • Study Protocol (2012-01-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT01462253/Prot_001.pdf